CLINICAL TRIAL: NCT06667453
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of PGN-EDODM1 in Adult Participants With Myotonic Dystrophy Type 1 (FREEDOM2-DM1)
Brief Title: A Clinical Study of PGN-EDODM1 in People With Myotonic Dystrophy Type 1
Acronym: FREEDOM2-DM1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PepGen Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGN-EDODM1-102
Record Dates: First submitted 2024-10-22; First posted 2024-10-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Myotonic Dystrophy 1
Keywords: DM1; Myotonic Dystrophy 1; Myotonic Dystrophy; PepGen; PGN-EDODM1; Myotonic Muscular Dystrophy; Steinert's Disease
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PGN-EDODM1 (Experimental): Participants will be randomized to receive ascending doses of PGN-EDODM1, once every 4 weeks (Q4W) for 12 weeks
  Interventions: Drug: PGN-EDODM1
- Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive doses of saline (0.9% NaCl), once every 4 weeks (Q4W) for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PGN-EDODM1 — Administered by intravenous (IV) infusion
  Arms: PGN-EDODM1
Other: Placebo — Administered by intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about the effects of an investigational medicine, PGN-EDODM1, to see how safe and tolerable multiple administrations of PGN-EDODM1 are for people with myotonic dystrophy type 1 (DM1) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DM1, as defined as having a repeat sequence in the DMPK gene with at least 100 CTG repeats
* Medical Research Council (MRC) score of ≥ Grade 4- in bilateral tibialis anterior (TA) muscles (the ability to move through full range of motion and hold against at least moderate pressure from the examiner)
* Presence of myotonia
* Body Mass Index (BMI) of < 32.0 kg/m^2

Exclusion Criteria:

* Congenital DM1
* Known history or presence of any clinically significant conditions that may interfere with study safety assessments
* Abnormal laboratory tests at screening considered clinically significant by the Investigator
* Medications specific for the treatment of myotonia within 2 weeks prior to screening
* Percent predicted forced vital capacity (FVC) <40%
* Use of an investigational drug, device, or product within 30 days of 5 half-lives of the study drug (whichever is longer) prior to Screening

Note: Other inclusion and exclusion criteria may apply.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by number of participants with Adverse Events (AEs) | Baseline through Day 112

SECONDARY OUTCOMES:
Maximum Observed Plasma Drug Concentration (Cmax) of PGN-EDODM1 | Day 1 through Day 84
Time to Maximum Observed Plasma Drug Concentration (Tmax) of PGN-EDODM1 | Day 1 through Day 84
Apparent Terminal Half-Life (t½) of PGN-EDODM1 | Day 1 through Day 84
Area Under the Concentration-time Curve of PGN-EDODM1 | Day 1 through Day 84
Change in splicing index in skeletal muscle tissue | Baseline through Day 91
Change in myotonia as measured by video Hand Opening Time (vHOT) | Baseline through Day 112
Hand grip strength | Baseline through Day 112
  by dynamometer
Change in mobility as measured by 10 meter walk/run time | Baseline through Day 112

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - Ottawa Hospital Research Institute (OHRI), Ottawa, Ontario
  - CIUSSS du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Montreal Neurological Institute, Montreal, Quebec
- United Kingdom (3):
  - Salford Royal Hospital, Salford, England
  - University College London Hospitals NHS Foundation Trust, London, UK
  - Newcastle Upon Tyne Hospitals, Newcastle upon Tyne